CLINICAL TRIAL: NCT05868577
Title: Infracalcaneal Peppering Injection Technique for Chronic Plantar Fasciitis: Protocol for a Parallel Randomized Clinical Trial
Brief Title: Infracalcaneal Peppering Injection Technique for Chronic Plantar Fasciitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00095622; UL1TR001420 (NIH)
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2024-03

CONDITIONS: Chronic Plantar Fasciitis
Keywords: corticosteroid injection; infracalcaneal peppering injection; Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Adrenal Cortex Hormones; Craniospinal Irradiation; Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: All patients ages 18 years and up with a diagnosis of plantar heel pain will be screened for inclusion into the study.
Who Masked: Participant, Investigator
Masking Description: A nurse or staff member will open a previously prepared and sealed opaque envelope (prepared beforehand by the clinical coordinator) labeled with the participant identification (ID) of the patient, which will be unique to the individual and different from their Medical Record Number (MRN). In this envelope, they will discover the patient's assigned treatment arm. The nurse or staff member will then prepare the syringe with the assigned treatment arm. Once the syringe is filled with the designated substance, the syringe will be wrapped with opaque tape or dark Coban wrap to conceal the contents in the syringe for both the PI and study participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- corticosteroid injection/ local anesthetic (CSI/LA) (Experimental): The PI will then administer the (CSI/LA) injection using an infracalcaneal needle peppering technique as follows:
  1. The hypodermic needle is inserted using infracalcaneal injection approach.
  2. The hypodermic needle is withdrawn while at the same depositing injectate
  3. The hypodermic needle is redirected without emerging from the skin. The PI will perform steps 1-3 standardly 20-25 times.
  Interventions: Drug: Corticosteroid injection (CSI) with local anesthetic (LA)
- local anesthetic (LA)/Saline injection (Placebo Comparator): The PI will then administer the (LA/Saline) injection using an infracalcaneal needle peppering technique as follows:
  1. The hypodermic needle is inserted using infracalcaneal injection approach.
  2. The hypodermic needle is withdrawn while at the same depositing injectate
  3. The hypodermic needle is redirected without emerging from the skin. The PI will perform steps 1-3 standardly 20-25 times.
  Interventions: Drug: Local anesthetic (LA) with Saline injection

INTERVENTIONS:
Drug: Corticosteroid injection (CSI) with local anesthetic (LA) — The PI will then administer the injection using an infracalcaneal needle peppering
  Other Names: Corticosteroid injection
  Arms: corticosteroid injection/ local anesthetic (CSI/LA)
Drug: Local anesthetic (LA) with Saline injection — The PI will then administer the injection using an infracalcaneal needle peppering
  Other Names: Local anesthetic injection
  Arms: local anesthetic (LA)/Saline injection

SUMMARY:
Although no single treatment has shown superiority, short-term pain relief may be offered via a targeted local corticosteroid injection (CSI), used often in combination with local anesthetic (LA), which may reduce plantar fasciitis symptoms for up to 1 month. Moreover, administering a CSI is relatively quick and easy for any Provider to perform, though it is not without potential deleterious side effects and risks, including fibroblast degradation, fat pad atrophy, skin depigmentation, and even plantar fascia rupture.

DETAILED DESCRIPTION:
Research performed in other musculoskeletal disorders (e.g. lateral epicondylitis) suggest that the "method" (i.e peppering vs single bolus deposition) of injection is more favorable than the steroid itself, though evidence for this positive effect in plantar fasciitis is rather scarce.

Injection via peppering is a minimally invasive percutaneous technique which involves repeatedly fenestrating the pathologic site (i.e. plantar fascia) via hypodermic needle insertion at the tender area, then sequentially injecting a substance, withdrawing, redirecting, and reinserting all without emerging from the skin. Though hypothetical, this technique is thought to disrupt the degenerative process of Plantar Fasciitis (PF), encouraging both localized bleeding and fibroblastic proliferation and stimulating a local inflammatory response that would trigger the body's own reparative mechanism, leading to recovery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older
* Patient reported history of plantar heel pain and confirmed clinical tenderness of pain with direct palpation of the medial calcaneal tubercle on baseline exam
* Diagnosis of chronic plantar fasciitis, defined for study purposes as symptoms greater than or equal to 6 weeks in duration

Exclusion Criteria:

* Individuals less than 18 years of age
* Pregnancy
* History of receiving a local heel injection (i.e. corticosteroid injection (CSI) or other injectate) within the last 3 months
* Prior heel trauma or surgery
* Allergy to local corticosteroid or local anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Jones, DPM, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Corticosteroid Injection/ Local Anesthetic (CSI/LA): The PI will then administer the (CSI/LA) injection using an infracalcaneal needle peppering technique as follows:
  1. The hypodermic needle is inserted using infracalcaneal injection approach.
  2. The hypodermic needle is withdrawn while at the same depositing injectate
  3. The hypodermic needle is redirected without emerging from the skin. The PI will perform steps 1-3 standardly 20-25 times.
  Corticosteroid injection (CSI) with local anesthetic (LA): The PI will then administer the injection using an infracalcaneal needle peppering
- Local Anesthetic (LA)/Saline Injection: The PI will then administer the (LA/Saline) injection using an infracalcaneal needle peppering technique as follows:
  1. The hypodermic needle is inserted using infracalcaneal injection approach.
  2. The hypodermic needle is withdrawn while at the same depositing injectate
  3. The hypodermic needle is redirected without emerging from the skin. The PI will perform steps 1-3 standardly 20-25 times.
  Local anesthetic (LA) with Saline injection: The PI will then administer the injection using an infracalcaneal needle peppering
Period: Overall Study
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Started | 21 | 20
Completed | 16 | 15
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12.4) | 53.5 (13.1) | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 19 | 16 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Diabetes Mellitus Diagnosis [Number; unit: participants] | 4 | 1 | 5
Clinical Duration of Symptoms [Mean (Standard Deviation); unit: days] | 205 (323) | 125 (217) | 166 (272.5)
Plantar Fascia Thickness [Mean (Standard Deviation); unit: mm] | 5.1 (1.7) | 5.2 (2.8) | 5.2 (1.4)
Heel Spur Size [Mean (Standard Deviation); unit: mm] | 5.1 (3.3) | 5.1 (3.9) | 5.1 (3.5)
Patients Diagnosed with Heel Spur [Number; unit: participants] | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Score - General Heel Tenderness
Description: A sheet of paper with a printed VAS scale will be given to the patient. The patient will be instructed to make a bold dot on the line based on how they rate their general heel pain, using the parameters listed on the scale (0 meaning no pain, 20 meaning mild pain, 50 meaning moderate pain, 80 meaning extreme pain, and 100 meaning the worst pain imaginable). Range 0-100.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 21 | 20
score on a scale | 46.7 (19.3) | 47.5 (17.7)

2. Primary Outcome: Visual Analog Scale Score - General Heel Tenderness
Description: A sheet of paper with a printed visual analog score scale will be given to the patient. The patient will be instructed to make a bold dot on the line based on how they rate their general heel pain, using the parameters listed on the scale (0 meaning no pain, 20 meaning mild pain, 50 meaning moderate pain, 80 meaning extreme pain, and 100 meaning the worst pain imaginable). Range = 0-100.
Time Frame: Week 2
Population: For CSI/LA arm, 2 participants did not complete the study, 2 participant missed Week 2 appointment. For LA/saline arm, 2 participants missed Week 2 appointment, 1 participant did not complete the study, 2 missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 17 | 15
score on a scale | 35.9 (23.1) | 41.8 (20.3)

3. Primary Outcome: Visual Analog Scale Score - General Heel Tenderness
Description: A sheet of paper with a printed visual analog scale will be given to the patient. The patient will be instructed to make a bold dot on the line based on how they rate their general heel pain, using the parameters listed on the scale (0 meaning no pain, 20 meaning mild pain, 50 meaning moderate pain, 80 meaning extreme pain, and 100 meaning the worst pain imaginable). Range 0-100.
Time Frame: Week 4
Population: For CSI/LA arm, 2 participant missed Week 4 appointment, 2 participants did not complete the study 1 missing data. For LA/saline arm, 3 missed appointment, 1 participants did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 16 | 16
score on a scale | 36.6 (25.6) | 32.6 (21.8)

4. Primary Outcome: Visual Analog Scale Score - General Heel Tenderness
Description: A sheet of paper with a printed visual analog scale will be given to the patient. The patient will be instructed to make a bold dot on the line based on how they rate their general heel pain, using the parameters listed on the scale (0 meaning no pain, 20 meaning mild pain, 50 meaning moderate pain, 80 meaning extreme pain, and 100 meaning the worst pain imaginable). Range = 0-100.
Time Frame: Week 8
Population: For the CSI.LA arm, 4 participants did not complete the study, 1 participant did not have this data point collected at Week 8 appointment, and 3 participants missed Week 8 appointment. For the LA/saline arm, 4 patients did not complete the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 13 | 16
score on a scale | 29.3 (30.8) | 22.6 (19.6)

5. Primary Outcome: Visual Analog Scale Score - General Heel Tenderness
Description: as for outcome 4
Time Frame: Week 12
Population: For CSI/LA arm, 5 participants did not complete the study. For LA/saline arm, 4 patients did not complete the study, and 1 patient missed Week 12 appointment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 16 | 15
score on a scale | 31.4 (25.3) | 24.4 (23.7)

6. Primary Outcome: Visual Analog Scale Score - First Step Pain
Description: A sheet of paper with a printed visual analog scale will be given to the patient. The patient will be instructed to make a bold dot on the line based on how they rate their first step heel pain, using the parameters listed on the scale (0 meaning no pain, 20 meaning mild pain, 50 meaning moderate pain, 80 meaning extreme pain, and 100 meaning the worst pain imaginable). Range = 0-100.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 21 | 20
score on a scale | 62.6 (20.2) | 70.6 (15.3)

7. Primary Outcome: Visual Analog Scale Score - First Step Pain
Description: as for outcome 6
Time Frame: Week 2
Population: For the CSI/LA arm, 2 participants did not complete the study, 2 person missed Week 2 appointment. For LA/saline arm, 2 participants missed Week 2 appointment, 1 participant did not complete study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 17 | 17
score on a scale | 40.4 (26.3) | 50.6 (23.1)

8. Primary Outcome: Visual Analog Scale Score - First Step Pain
Description: as for outcome 6
Time Frame: Week 4
Population: For the CSI/LA arm, 2 participants missed Week 4 appointment, 2 participants did not complete study. For LA/saline injection arm, 3 participants did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 17 | 17
score on a scale | 40.3 (27.9) | 37.8 (23.6)

9. Primary Outcome: Visual Analog Scale Score - First Step Pain
Description: as for outcome 6
Time Frame: Week 8
Population: For the CSI/LA arm, 4 participants did not complete the study, 3 participants missed Week 8 appointment. For the LA/saline arm, 1 participant did not have this data point collected, 4 participants did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 14 | 15
score on a scale | 38.7 (32.7) | 24.9 (23.0)

10. Primary Outcome: Visual Analog Scale Score - First Step Pain
Description: as for outcome 6
Time Frame: Week 12
Population: For the CSI/LA arm, 5 participants did not complete study. For the LA/saline arm, 4 participants did not complete the study, 1 participant missed Week 12 appointment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 16 | 15
score on a scale | 37.1 (29.8) | 22.9 (22.6)

11. Primary Outcome: Foot Function Index (FFI) Score
Description: Questionnaire that measures pain, activity limitation, and disability in the foot. The FFI consists of 23 items grouped into three subscales: (1) Pain (9 items); (2) Disability (9 items); and (3) Activity Limitation (5 items). Each item is rated on a scale from 0-9 for the Pain and Disability subscales and 0-5 for the Activity Limitation subscale. For each subscale, scores are summed, divided by the maximum possible total for applicable items (excluding any marked "not applicable"), and multiplied by 100 to yield a percentage score from 0 to 100. Lower FFI scores indicate better foot function, while higher FFI scores reflect greater impairment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 21 | 20
score on a scale | 42.4 (13.5) | 43.5 (15.2)

12. Primary Outcome: Foot Function Index (FFI) Score
Description: as for outcome 11
Time Frame: Week 2
Population: For the CSI/LA arm, 2 participants did not complete study, 1 missed appointment. For LA/saline arm, 1 participant missed Week 2 appointment, 1 participant did not complete study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 18 | 18
score on a scale | 28.3 (16.6) | 33.1 (15.5)

13. Primary Outcome: Foot Function Index (FFI) Score
Description: as for outcome 11
Time Frame: Week 4
Population: For CSI/LA arm, 1 participant missed Week 4 appointment, 2 participants did not complete study. For the LA/saline arm, 3 participants did not complete study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 18 | 17
score on a scale | 22.2 (16.9) | 25.3 (18.8)

14. Primary Outcome: Foot Function Index (FFI) Score
Description: as for outcome 11
Time Frame: Week 8
Population: For the CSI/LA arm, 3 participants missed Week 8 appointment, 4 participants did not finish study. For the LA/saline arm, 4 participants did not finish study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 14 | 16
score on a scale | 22.6 (20.2) | 17.1 (17.2)

15. Primary Outcome: Foot Function Index (FFI) Score
Description: as for outcome 11
Time Frame: Week 12
Population: For the CSI/LA arm, 5 participants did not complete study. For the LA/saline arm, 5 participants did not complete study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 16 | 15
score on a scale | 26.5 (23.3) | 18.6 (20.2)

16. Secondary Outcome: Exit Survey Score
Description: Upon completion of study related procedures and assessments, participants will be given a paper exit survey to complete. 5 questions asked relating to their experience in the study and if they would recommend the study to others. Total score range 1-10 with 1 being worst experience and 10 being best experience.
Time Frame: Week 12
Population: For the CSI/LA arm, 5 participants did not complete the study, 1 missing data. For the LA/saline arm, 5 did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 15 | 15
score on a scale | 8.8 (1.8) | 9.6 (0.7)

17. Secondary Outcome: Number of Completed Exercises
Description: Participants will document in a daily exercise diary if any of the three recommended exercises (calf stretching, plantar fascia specific stretching, and loading exercise) were completed. Participants will also be asked to document why exercises were not completed if applicable.
Time Frame: Week 2, Week 4, Week 8, and Week 12
Population: W2: CSI/LA 2 didn't complete study, 2 missed appt, 3 no diary; LA/saline 1 didn't complete study, 1 missed appt, 2 no diary. W4: CSI/LA 3 no diary, 1 missed appt, 2 didn't complete study; LA/saline 3 no diary, 3 didn't complete study. W8: CSI/LA, 1 no diary, 4 didn't complete study, 3 missed appt; LA/saline 4 didn't finish study, 1 no diary. W12: CSI/LA 5 no diary, 5 didn't finish study; LA/saline 4 no diary, 5 didn't complete study.
Measure: Mean (Standard Deviation); unit: exercises completed
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 21 | 20
exercises completed
  week 2: number analyzed (Participants) | 14 | 16
  week 2 | 14.1 (3.0) | 13.8 (1.3)
  week 4: number analyzed (Participants) | 15 | 14
  week 4 | 13.8 (2.7) | 15.9 (3.3)
  week 8: number analyzed (Participants) | 13 | 15
  week 8 | 26.2 (4.9) | 25.1 (5.6)
  week 12: number analyzed (Participants) | 11 | 11
  week 12 | 26.9 (4.2) | 27.2 (3.4)

18. Secondary Outcome: Heel Pressure Threshold Score - Symptomatic Foot
Description: Using a dolorimeter each participant's heel pressure threshold will be assessed. Level of pain on a 35-point scale will be noted with 0 meaning no pain and 35 meaning extreme pain.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: Baseline: CSI/LA 1 outlier, data excluded. W2: CSI/LA 2 didn't complete study, 2 missed appt; LA/saline 1 didn't complete study, 3 missed appt. W4: CSI/LA 2 missed appt, 2 didn't complete study; LA/saline 3 didn't complete study. W8: CSI/LA 4 didn't complete study, 5 missed appt; LA/saline 4 didn't finish study, 1 missing data, 2 outliers data excluded. W12: CSI/LA 5 didn't finish study, 1 missing data; LA/saline 5 didn't complete study, 1 missing data, 2 outliers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 21 | 20
score on a scale
  baseline: number analyzed (Participants) | 20 | 20
  baseline | 12.3 (7.2) | 12.3 (6.8)
  week 2: number analyzed (Participants) | 17 | 16
  week 2 | 12.6 (6.8) | 12.8 (6.0)
  week 4: number analyzed (Participants) | 17 | 17
  week 4 | 12.5 (5.7) | 14.1 (5.9)
  week 8: number analyzed (Participants) | 12 | 13
  week 8 | 13.4 (6.8) | 13.1 (5.9)
  week 12: number analyzed (Participants) | 15 | 12
  week 12 | 12.8 (7.0) | 15.4 (7.7)

19. Secondary Outcome: Heel Pressure Threshold Score - Asymptomatic Foot
Description: as for outcome 18
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: BL:CSI/LA 1 outlier data excluded; LS/saline 3 outliers. W2:CSI/LA 2 didn't complete study, 2 missed appt; LA/saline 1 didn't complete study, 3 missed appt, 2 outliers. W4:CSI/LA 2 missed appt, 2 didn't complete study; LA/saline 3 didn't complete study, 3 outliers. W8:CSI/LA 4 didn't complete study, 5 missed appt; LA/saline 4 didn't finish study, 1 missing data, 4 outliers. W12:CSI/LA 5 didn't finish study, 1 missing; LA/saline 5 didn't complete study, 1 missed appt, 4 outliers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 21 | 20
score on a scale
  baseline: number analyzed (Participants) | 20 | 17
  baseline | 16.0 (6.5) | 18.0 (11.5)
  week 2: number analyzed (Participants) | 17 | 14
  week 2 | 15.7 (7.7) | 19.2 (12.1)
  week 4: number analyzed (Participants) | 17 | 14
  week 4 | 14.5 (5.3) | 17.1 (8.7)
  week 8: number analyzed (Participants) | 12 | 11
  week 8 | 15.6 (6.8) | 15.4 (5.4)
  week 12: number analyzed (Participants) | 15 | 10
  week 12 | 14.4 (6.1) | 15.2 (5.9)

20. Secondary Outcome: Heel Tenderness Score - Symptomatic Foot
Description: The physician will assess heel pain on palpation. Heel tenderness index will be used which has a range of 0-3 points (0 points = no pain, 1 point = painful, 2 points = painful and winces, 3 points = painful, winces, and withdraws).
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: WK 2: CSI/LA 2 missed appt, 2 did not complete study; LA/saline 3 missed appt, 1 did not complete study. WK 4: CSI/LA 2 missed appt, 2 did not finish study; LA/saline 3 did not finish study. WK 8: CSI/LA 5 missed appt, 4 did not finish study; LA/saline 4 did not finish study, 1 missed appt. WK 12: CSI/LA 1 missed data, 5 did not finish study; LA/saline 5 did not finish study, 1 missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 21 | 20
score on a scale
  baseline | 1.95 (0.65) | 1.75 (0.62)
  week 2: number analyzed (Participants) | 17 | 16
  week 2 | 1.29 (0.57) | 1.38 (0.60)
  week 4: number analyzed (Participants) | 17 | 17
  week 4 | 1.18 (0.78) | 1.35 (0.76)
  week 8: number analyzed (Participants) | 12 | 15
  week 8 | 1.7 (0.55) | 1.13 (0.72)
  week 12: number analyzed (Participants) | 15 | 14
  week 12 | 1.0 (0.82) | 1.0 (1.0)

21. Secondary Outcome: Heel Tenderness Score - Asymptomatic Foot
Description: as for outcome 20
Time Frame: Baseline, week 2, week 4, week 8, week 12
Population: Baseline: CSI/LA 2 missing data; LA/saline 2 missing data. WK 2: CSI/LA 2 missed appt, 2 did not complete study; LA/saline 1 did not complete study, 3 missed appt, 2 missing data. WK 4: CSI/LA 2 missed appt, 2 did not finish study; LA/saline 3 did not finish study. WK 8: CSI/LA 5 missed appt, 4 did not finish study; LA/saline 4 did not finish study, 1 missed appointment. WK 12: CSI/LA 1 missed data, 5 did not finish study; LA/saline 1 missing data, 5 did not finish study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
Number analyzed (Participants) | 21 | 20
score on a scale
  baseline: number analyzed (Participants) | 19 | 18
  baseline | 0.32 (0.57) | 0.33 (0.58)
  week 2: number analyzed (Participants) | 17 | 14
  week 2 | 0.18 (0.38) | 0.21 (0.56)
  week 4: number analyzed (Participants) | 17 | 17
  week 4 | 0 (0) | 0.12 (0.47)
  week 8: number analyzed (Participants) | 12 | 15
  week 8 | 0 (0) | 0.07 (0.25)
  week 12: number analyzed (Participants) | 15 | 14
  week 12 | 0.27 (0.57) | 0.21 (0.77)

ADVERSE EVENTS:
Time Frame: Baseline through Week 12
Arm/Group | Corticosteroid Injection/ Local Anesthetic (CSI/LA) | Local Anesthetic (LA)/Saline Injection
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 2/21 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroid Injection/ Local Anesthetic (CSI/LA) (N=21) | Local Anesthetic (LA)/Saline Injection (N=20)
Fall (General disorders) | 2 (2) | 0 (0)
oral surgery (General disorders) | 0 (0) | 1 (1)
mass with sensation (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT05868577/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT05868577/ICF_002.pdf